CLINICAL TRIAL: NCT03035474
Title: Care Optimization Through Patient and Hospital Engagement Clinical Trial for Heart Failure (CONNECT-HF)
Brief Title: Care Optimization Through Patient and Hospital Engagement Clinical Trial for Heart Failure
Acronym: CONNECT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Pro00074513
Record Dates: First submitted 2017-01-05; First posted 2017-01-30 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Quality Improvement
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct & Digital (Other): Health system engagement to improve local QI programs and patient engagement to improve self-management/medication adherence
  Interventions: Other: Digital Engagement; Other: Direct Engagement
- Direct & Registry (Other): Health system engagement to improve local QI programs and patient and control
  Interventions: Other: Direct Engagement
- Digital & Registry (Other): Patient engagement to improve self-management/medication adherence and control
  Interventions: Other: Digital Engagement
- Registry (No Intervention): Control

INTERVENTIONS:
Other: Digital Engagement — Patient engagement to improve self-management/medication adherence
  Arms: Digital & Registry; Direct & Digital
Other: Direct Engagement — Health system engagement to improve local QI programs
  Arms: Direct & Digital; Direct & Registry

SUMMARY:
CONNECT-HF is a large-scale, pragmatic, cluster-randomized clinical trial to evaluate the effect of a customized, multifaceted, health system-level quality-improvement (QI) program compared with usual care on heart failure (HF) outcomes and HF quality-of-care metrics.

DETAILED DESCRIPTION:
This trial will be a large-scale, pragmatic, cluster-randomized clinical trial to evaluate the effect of a customized, multifaceted, health system-level quality-improvement (QI) program compared with usual care on heart failure (HF) outcomes and HF quality-of-care metrics. Outcomes will be assessed following discharge for participants hospitalized with acute HF and reduced left ventricular ejection fraction. All participants in the trial will be consented for follow-up as part of the CONNECT-HF registry on clinical outcomes, medication use, and participant-centered outcomes, including quality-of-life (QOL) assessments will be collected up to 12 months post-discharge at pre-specified intervals (6 weeks and 3, 6, and 12 months).

The health-system QI program will involve site visits and ongoing mentoring from teams of healthcare professionals with specialized training and field experience to help health systems and individual hospitals to design local QI plans.

A key substudy will assess a participant-engagement strategy (digital) of a mobile application utilizing behavioral tools to reinforce health behaviors, including self-monitoring/self-management and medication adherence.

Follow-up will occur via a centralized telephone interview by trained personnel via the DCRI Call Center. At each interview, participants will be asked to report current medications, rehospitalizations, and QOL assessments. Based on participant-reported events, medical billing data for rehospitalizations, emergency department visits, and procedures will be obtained.

Quality of life assessments will include the Kansas City Cardiomyopathy Questionnaire (KCCQ) and EuroQOL five dimensions questionnaire (EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute HF as a primary cause of hospitalization

  * Hospitalizations for acute HF will be determined by local clinician-investigators but should include the following:
  * Symptoms (eg, dyspnea, fatigue), signs (eg, elevated jugular venous pressure, peripheral edema), or laboratory/imaging evidence of HF (eg, pulmonary congestion on chest x-ray, elevated natriuretic peptide levels) during the hospitalization and
  * Treatments aimed at acute HF (eg, intravenous diuretics, vasodilators, or inotropes)
* LVEF ≤ 40% based on last local measurement using echocardiography, multigated acquisition scan, computed tomography (CT) scanning, magnetic resonance imaging, or ventricular angiography
* Planned discharge to home or other supported care facility where patients are individually responsible for medication management

Exclusion Criteria:

* Prior heart transplant or current/planned left ventricular assistance device
* Chronic kidney disease requiring dialysis
* Terminal illness other than HF, such as malignancy, or with a life expectancy of less than 1 year as determined by the enrolling clinician-investigator
* Unable to participate in longitudinal follow-up, such as plans to move outside the US in the following year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5749 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Time-to-first HF rehospitalization or death during the 12-months post-discharge | 12-months after discharge
Improvement in an opportunity-based composite score of adherence to quality metrics for HF. | Baseline to 12 months post discharge
  The opportunity-based composite score will be created to grade the quality of care provided. The numerator will be the number of times that good care is provided; the denominator will be the number of opportunities available. The score will consist of the following quality metrics assessed at the time of hospital discharge and during outpatient follow-up:
  * Use of evidence-based specific β-blockers at ≥ 50% target dose
  * ACE-I, ARB, or sacubitril/valsartan use at ≥ 50% target dose
  * Aldosterone antagonist use
  * Anticoagulation use in participants with atrial fibrillation
  * In participants with an LVEF ≤ 35%, implantable cardioverter defibrillator placement including cardiac resynchronization therapy placement for participants with sinus rhythm, LBBB, and a QRS ≥ 150 ms
  * Attendance at 1 or more of the following: a multidisciplinary HF disease management program, a cardiac rehabilitation program, or HF group educational classes

SECONDARY OUTCOMES:
Improvement in an opportunity-based composite score for adherence to HF discharge quality measures | Baseline through study completion, an average of 3 years
  The opportunity-based composite score will be created to grade the quality of care provided. The numerator will be adherence to medications; the denominator will be the number of opportunities available. The per-opportunity adherence rate will consist of the following quality metrics assessed at the time of hospital discharge:
  * ACE-I, ARB, or sacubitril/valsartan prescription at discharge
  * ß-blocker prescription at discharge
  * Discharge instructions addressing activity level, diet, discharge medications, follow-up appointment, weight monitoring, and how to respond to a change in symptoms
  * LVEF assessment
  * Smoking cessation counseling
  * Medication adherence
If there is a significant positive effect on at least one of the primary endpoints, then participant-level healthcare expenditures | 6 months and 1 year postdischarge
Cumulative number of primary composite events of death and total (first and recurrent) HF hospitalizations | Baseline through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Adam DeVore, MD, MHS, Principal Investigator — Duke University
Locations (154):
- United States (154):
  - University of Alabama Hospital, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Arkansas Heart Hospital and Clinics, Little Rock, Arkansas
  - San Gorgonio Memorial Hospital, Banning, California
  - Memorial Medical Center, Modesto, California
  - Dignity Health Sequoia Hospital, Redwood City, California
  - Riverside Community Hospital, Riverside, California
  - Sutter Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - UC Health Memorial, Colorado Springs, Colorado
  - Northern Colorado Medical Center, Greeley, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - JFK Medical Center, Atlantis, Florida
  - Manatee Memorial Hospital, Bradenton, Florida
  - Blake Medical Center, Bradenton, Florida
  - Broward Health Imperial Point, Fort Lauderdale, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Baptist Hospital, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - South Miami Hospital, South Miami, Florida
  - Bayfront Health - St. Petersburg, St. Petersburg, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - AU Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center, Navicent Health (THE), Macon, Georgia
  - The Queens Medical Center, Honolulu, Hawaii
  - Copley Memorial Hospital, Aurora, Illinois
  - Presence Mercy Medical Center, Aurora, Illinois
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - Specialty Physicians of Illinois, Olympia Fields, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - St Johns Hospital, Springfield, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Indiana University Health Bloomington, Bloomington, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Reid Health, Richmond, Indiana
  - Genesis Medical Center-Davenport, Davenport, Iowa
  - King's Daughters Medical Center, Ashland, Kentucky
  - KentuckyOne Health - Saint Joseph Hospital, Lexington, Kentucky
  - Norton Women and Children's Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Baptist Health Madisonville, Madisonville, Kentucky
  - Rapides Regional Medical Center, Alexandria, Louisiana
  - Natchitoches Regional Medical Center, Natchitoches, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Louisiana State University-Health Science Center- Shreveport, Shreveport, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Adventist HealthCare Shady Grove, Rockville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Code Hospital, Hyannis, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - St. John Macomb-Oakland, Madison Heights, Michigan
  - MidMichigan Medical Center Midland, Midland, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - McLaren - Northern Michigan, Petoskey, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - St Lukes Hospital, Duluth, Minnesota
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - St. Mary's Medical Center, Blue Springs, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - Billings Clinic Hospital, Billings, Montana
  - Glacier View Research Institute-Cardiology, Kalispell, Montana
  - Bryan Medical Center, Lincoln, Nebraska
  - University Medical Center, Las Vegas, Nevada
  - Southern NH Medical Center, Nashua, New Hampshire
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - St. Peter's Hospital, Albany, New York
  - Huntington Hospital, Huntington, New York
  - United Health Services Hospitals, Johnson City, New York
  - Mount Sinai Beth Israel, New York, New York
  - Ellis Hospital, Schenectady, New York
  - Staten Island University Hospital, Staten Island, New York
  - Richmond University Medical Center, Staten Island, New York
  - University Hospital (Stony Brook), Stony Brook, New York
  - St. Joseph's Hospital, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Charlotte-Mecklenburg Hospital Authority, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Duke Cardiology of Lumberton, Lumberton, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - WakeMed, Raleigh, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - Summa Health, Akron, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University Hospitals - Elyria Medical Center, Elyria, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - OHSU Hospital and Clinics, Portland, Oregon
  - Memorial Medical Center, Johnstown, Pennsylvania
  - WellSpan Good Samaritan Hospital, Lebanon, Pennsylvania
  - Self Regional Healthcare, Greenwood, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Christus Good Shepherd Medical Center, Longview, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Hospital, San Antonio, Texas
  - Guadalupe Regional Medical Center, Seguin, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - CJW Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Wheeling Hospital, Wheeling, West Virginia
  - Mayo Clinic Health System Franciscan Medical Center, La Crosse, Wisconsin
  - Ascension Columbia St. Mary's Hospital, Milwaukee, Wisconsin
  - Ascension-All Saints, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao VN, Kaltenbach LA, Granger BB, Fonarow GC, Al-Khalidi HR, Albert NM, Butler J, Allen LA, Lanfear DE, Ariely D, Miller JM, Brodsky MA, Lalonde TA, Lafferty JC, Granger CB, Hernandez AF, Devore AD; Durham, North Carolina; Los Angeles, California; Cleveland, Ohio; Jackson, Misssissippi, Aurora, Colorado; Detroit, Michigan; Ewa Beach, Hawaii; Staten Island, New York. The Association of Digital Health Application Use With Heart Failure Care and Outcomes: Insights From CONNECT-HF. J Card Fail. 2022 Oct;28(10):1487-1496. doi: 10.1016/j.cardfail.2022.07.050. Epub 2022 Jul 26. PMID 35905867
- [Derived] DeVore AD, Granger BB, Fonarow GC, Al-Khalidi HR, Albert NM, Lewis EF, Butler J, Pina IL, Allen LA, Yancy CW, Cooper LB, Felker GM, Kaltenbach LA, McRae AT, Lanfear DE, Harrison RW, Disch M, Ariely D, Miller JM, Granger CB, Hernandez AF. Effect of a Hospital and Postdischarge Quality Improvement Intervention on Clinical Outcomes and Quality of Care for Patients With Heart Failure With Reduced Ejection Fraction: The CONNECT-HF Randomized Clinical Trial. JAMA. 2021 Jul 27;326(4):314-323. doi: 10.1001/jama.2021.8844. PMID 34313687
- [Derived] DeVore AD, Granger BB, Fonarow GC, Al-Khalidi HR, Albert NM, Lewis EF, Butler J, Pina IL, Heidenreich PA, Allen LA, Yancy CW, Cooper LB, Felker GM, Kaltenbach LA, McRae AT, Lanfear DE, Harrison RW, Kociol RD, Disch M, Ariely D, Miller JM, Granger CB, Hernandez AF. Care Optimization Through Patient and Hospital Engagement Clinical Trial for Heart Failure: Rationale and design of CONNECT-HF. Am Heart J. 2020 Feb;220:41-50. doi: 10.1016/j.ahj.2019.09.012. Epub 2019 Oct 23. PMID 31770656